CLINICAL TRIAL: NCT06154291
Title: Phase I/II, Multi Center, Open Label, First-in-human, Dose Escalation and Expansion Study to Investigate the Safety, Pharmacokinetics, and Anti-tumors Efficacy of the Glyco-humanized Polyclonal Antibody XON7 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: FIH XON7 in Advanced/Metastatic Solid Tumors
Acronym: FIPO23
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xenothera SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT 23-01; 2023-505266-29-00 (Other: EU CT number)
Record Dates: First submitted 2023-11-06; First posted 2023-12-04 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor; Metastatic Cancer
Keywords: Advanced or metastatic solid tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: The Part I component is a multicenter, open-label, multiple-dose, dose escalation, first-in-human study. Six dose levels are planned: 1.5; 3; 6; 12; 16 and 20mg/kg, Q2W (once every two weeks). Up to 45 participants with relapsed or refractory, advanced or metastatic solid tumors will be included.
  The Part II component is a multi-center, open-label, non-randomized, multi-cohorts, expansion trial with adaptive design.
  The selected cohorts of the study will investigate RP2D to determine the anti-tumors efficacy, safety, and tolerability of XON7 in participants with relapsed or refractory, advanced or metastatic solid tumors after failure to standard of care treatments.
  Up to 7 cohorts could be investigated. A maximum of 30 participants will be enrolled in each cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation part then Expansion part (Experimental): Dose Escalation part: Six dose levels are planned: 1.5; 3; 6; 12; 16 and 20mg/kg
  Expansion part: Up to 7 cohorts (1 cohort for one selected solid tumor type) could be investigated:
  Cohort E1: Non-small cell lung cancer (NSCLC) Cohort E2: Gastro-esophageal adenocarcinoma Cohort E3: Colorectal cancer (CRC) Cohort E4: Pancreatic cancer Cohort E5: Sarcoma Cohort E6: Triple-negative breast cancer (TNBC) Cohort E7: Ovarian cancer
  Interventions: Drug: XON7

INTERVENTIONS:
Drug: XON7 — The trial intervention (XON7) is a glyco-humanized polyclonal antibody drug which is formulated for intravenous (IV) administration

SUMMARY:
This is a two-stage trial consisting of a Part I, dose escalation and dose-finding component to establish the Maximal Tolerated Dose (MTD), if any, and Recommended Part 2 Dose (RP2D) of XON7, followed by a Part II component to investigate anti-tumors efficacy in selected solid tumor types and to further evaluate safety and tolerability of XON7 at RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed, written informed consent.
2. Male and female participant, age ≥ 18 years old (at the time consent is obtained)
3. Solid tumors indications:

   * Participant in phase I, must have a histologically or cytologically confirmed advanced or metastatic solid tumors for which no effective standard therapy is available. All tumor types except glioblastoma, could be included.
   * Participant in phase II, must have histologically or cytologically confirmed advanced or metastatic solid tumors of the following: NSCLC, gastro-esophageal adenocarcinoma, CRC, pancreatic cancer, Sarcoma, TNBC, or ovarian cancer.
4. Line of treatment: Participant must have solid tumors progressing after ≤ 4 lines of standard appropriate anticancer therapies for the specific tumor type, or for which the patient is ineligible. Participants whose cancers harbor molecular alterations for which targeted therapy is standard of care should have received health authority-approved appropriate targeted therapy for their tumor types before enrollment.
5. Measurable disease per RECIST version 1.1 - v5
6. (ECOG) performance status (PS) 0-1
7. Life expectancy of at least 12 weeks.
8. Adequate organ function
9. QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 msec or QTcF <480 msec for participants with bundle branch block.
10. In France, a participant will be eligible for inclusion in this trial only if either affiliated to or a beneficiary of a social security category.
11. Female participant who are not of child-bearing potential, and female participants of child-bearing potential who have a negative serum pregnancy test within 7 days prior to initial trial treatment. Female participants of child-bearing potential, and all male partners must consent to use a medically acceptable method of contraception throughout the trial period and for at least 60 days after the last dose of XON7. A barrier method of contraception must be included.
12. Male participant willing to use adequate contraceptive measures throughout the trial period and for at least 60 days after the last dose of trial intervention.
13. For phase II, participant in pharmacodynamics cohort must provide biopsy of a tumor lesion not previously irradiated during the screening period and must agree to provide at least one additional on-treatment biopsy between day 36 and 42 after trial intervention administration.
14. For phase II, participant in pharmacodynamics cohort must have accessible tumor tissue available for fresh biopsy except for ovarian cancer and sarcoma.

Exclusion Criteria:

1. A participant who has received more than 4 prior lines of therapy for advanced or metastatic disease.
2. A participant who has had a prior anti-cancer mAb within 3 weeks prior to trial Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier prior to trial Day 1.
3. A participant who has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to trial Day 1 or who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent (Except alopecia, hearing loss, grade 2 neuropathy or endocrinopathy managed with replacement therapy).
4. A participant with ≥Grade 3 toxicity related to prior immunotherapy leading to treatment discontinuation.
5. A participant whose toxicity related to prior treatment has not resolved to Grade 1 (except alopecia, hearing loss, grade 2 neuropathy or endocrinopathy managed with replacement therapy).
6. A participant who has received major surgery 2 weeks before the first dose of trial treatment or has not recovered adequately from the toxicity and/or complications from any surgery (major or minor) before initiating trial treatment.
7. Concomitant use of another experimental drug, or wash-out period of at least 5 half-lives for a previous experimental drug not completed before start of trial intervention
8. Participant treated with drugs known to prolong the QT interval
9. Participant with carcinomatous meningitis.
10. Central nervous system (CNS) metastases, with the exception of individuals who have been previously treated CNS metastases, are asymptomatic, and have had no requirement for steroids for 3 weeks prior to first dose of trial drug.
11. Malignancies other than disease under trial within 3 years prior to first dose of trial intervention.
12. History of autoimmune disease
13. Active or uncontrolled infections requiring systemic treatment (known human immunodeficiency virus infection, or positive test for hepatitis B surface antigen or hepatitis C).
14. Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the trial such as history or evidence of cardiovascular risk including any of the following:

    * Recent (within the past 6 months) history of serious uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities including second degree (Type II) or third-degree atrioventricular block.
    * Documented cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting, or bypass grafting within the past 6 months before enrollment.
    * Documented congestive heart failure (Class II, III, or IV) as defined by the New York Heart Association functional classification system (NYHA, 1994).
15. Prior allogeneic or autologous bone marrow transplantation or other solid organ transplantation.
16. Current active liver or biliary disease (Except for Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per investigator assessment).
17. Concurrent medical condition requiring the use of systemic immunosuppressive medications within 28 days before the first dose of trial treatment.
18. Recent history (within the past 6 months) of acute diverticulitis, inflammatory bowel disease, intra-abdominal abscess, or gastrointestinal obstruction.
19. Current or history of idiopathic pulmonary fibrosis, interstitial lung disease, or organizing pneumonia. Note: post-radiation changes in the lung related to prior radiotherapy and/or asymptomatic radiation-induced pneumonitis not requiring treatment may be permitted if agreed by the investigator and Medical Monitor.
20. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
21. Recent history (within 6 months) of uncontrolled symptomatic ascites or pleural effusions.
22. Participant who has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony- stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM- CSF], recombinant erythropoietin) within 2 weeks before the first dose of trial intervention.
23. Known, current drug or alcohol abuse.
24. Female participant who is pregnant or lactating.
25. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
26. Inability or unwillingness to comply with trial and/or follow-up procedures outlined in the protocol.
27. For France, patients under legal protection (safeguard, guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation part: Dose Limiting Toxicities (DLTs) | At the end of Cycle 1 (28 days)
  Investigator defined DLT during first treatment cycle
Dose Escalation part: treatment emergent adverse events (TEAEs) | At the end of Cycle 1 (28 days)
  An overall summary of AE occurrences with onset during the first treatment cycle will be presented; this will include the following AE attributes:
  * Preferred term,
  * Maximum CTCAE grade,
  * Outcome,
  * Time to first occurrence [days].
Dose Escalation part: clinically significant changes in Leucocytes count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Leucocytes Count (G/L)
Dose Escalation part: clinically significant changes in Red Blood Cells Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Red Blood Cells Count (T/L)
Dose Escalation part: clinically significant changes in Hemoglobin | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Hemoglobin (g/dL).
Dose Escalation part: clinically significant changes in Hematocrit | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Hematocrit (%).
Dose Escalation part: clinically significant changes in Absolute Neutrophil Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Absolute Neutrophil Count (G/L).
Dose Escalation part: clinically significant changes in Absolute Eosinophil Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Absolute Eosinophil Count (G/L).
Dose Escalation part: clinically significant changes in Absolute Basophil Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Absolute Basophil Count (G/L).
Dose Escalation part: clinically significant changes in Absolute Lymphocytes Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Absolute Lymphocytes Count (G/L).
Dose Escalation part: clinically significant changes in Absolute Monocytes Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Absolute Monocytes Count (G/L).
Dose Escalation part: clinically significant changes in Platelet Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Platelet Count (G/L).
Dose Escalation part: clinically significant changes in Albumin | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Albumin (g/L).
Dose Escalation part: clinically significant changes in Bicarbonate | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Bicarbonate (mmol/L).
Dose Escalation part: clinically significant changes in Total Bilirubin | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Total Bilirubin (µmol/L).
Dose Escalation part: clinically significant changes in Calcium | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Calcium (mmol/L).
Dose Escalation part: clinically significant changes in Urea | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Urea (mmol/L).
Dose Escalation part: clinically significant changes in Chloride | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Chloride (mmol/L).
Dose Escalation part: clinically significant changes in Creatinine | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Creatinine (µmol/L).
Dose Escalation part: clinically significant changes in Creatinine Clearance | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Creatinine Clearance (mL/min).
Dose Escalation part: clinically significant changes in Glucose | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Glucose (mmol/L).
Dose Escalation part: clinically significant changes in Magnesium | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Magnesium (mmol/L).
Dose Escalation part: clinically significant changes in Phosphate | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Phosphate (mmol/L).
Dose Escalation part: clinically significant changes in Potassium | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Potassium (mmol/L).
Dose Escalation part: clinically significant changes in Sodium | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Sodium (mmol/L).
Dose Escalation part: clinically significant changes in Total Protein | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Total Protein (g/L).
Dose Escalation part: clinically significant changes in Alanine aminotransferase (ALT) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Alanine aminotransferase (ALT) (U/L).
Dose Escalation part: clinically significant changes in Aspartate aminotransferase (AST) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Aspartate aminotransferase (AST) (U/L).
Dose Escalation part: clinically significant changes in Gamma-glutamyl transférase (GGT) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Gamma-glutamyl transférase (GGT) (U/L).
Dose Escalation part: clinically significant changes in Alkaline Phosphatase (ALP) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Alkaline Phosphatase (ALP) (U/L).
Dose Escalation part: clinically significant changes in Lactate dehydrogenase (LDH) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Lactate dehydrogenase (LDH) (U/L).
Dose Escalation part: clinically significant changes in Amylase | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Amylase (U/L).
Dose Escalation part: clinically significant changes in Lipase | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Lipase (U/L).
Dose Escalation part: clinically significant changes in Total Protein Creatine Kinase (CK) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Total Protein Creatine Kinase (CK) (U/L).
Dose Escalation part: clinically significant changes in Creatine kinase - cardiac muscle isoenzyme (CK-MB) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Creatine kinase - cardiac muscle isoenzyme (CK-MB) (U/L).
Dose Escalation part: clinically significant changes in Troponin T | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Troponin T (ng/L).
Dose Escalation part: clinically significant changes in Prothrombin Time (PT) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Prothrombin Time (PT) (Sec).
Dose Escalation part: clinically significant changes in INR (if under VKA Therapy) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in INR (if under VKA Therapy)
Dose Escalation part: clinically significant changes in Activated Partial Thromboplastin Time (aPTT) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Activated Partial Thromboplastin Time (aPTT) (Sec).
Dose Escalation part: clinically significant findings in blood pressure (BP) | At the end of Cycle 1 (28 days)
  Incidence and severity of clinically significant findings in blood pressure: Significant blood pressure increase will be defined as BP >150/100 mmHg in a subject without a history of hypertension or increased >20 mmHg (diastolic) from baseline measurement in a subject with a previous history of hypertension.
Dose Escalation part: clinically significant findings in electrocardiogram (ECGs) | At the end of Cycle 1 (28 days)
  Incidence of clinically significant findings in Electrocardiogram (ECG): Significant QTc prolongation will be defined as an interval ≥500 msec or an interval which increases by ≥60 msec over baseline
Expansion part: Anti-tumors efficacy | Within 3 months after XON7 initiation
  Objective response rate (ORR): defined as the proportion of participants with a confirmed complete response [CR] or confirmed partial response [PR] assessed by investigators according to RECIST v1.1.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of XON7 (Part 1): Cmax | Cycle 1-Day 1 Predose and Postdose: 5 minutes; 1; 2; 4; 8; 24; 72 or 96; 144 hours after the end of infusion. Cycle 1 Day 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 7 Day 1: Predose and 5 minutes after the end of infusion
  XON7 peak plasma concentration (Cmax) in plasma
Pharmacokinetics (PK) of XON7 (Part 2): Cmax | Cycle 1-Day 1; Cycle 2-Day 1; Cycle 3-Day 1; Cycle 6-Day 1; Cycle 9-Day1 and Cycle 12-Day 1: Predose and 5 minutes after the end of infusion
  XON7 peak plasma concentration (Cmax) in plasma
Pharmacokinetics (PK) of XON7 (Part 1): Tmax | Cycle 1-Day 1 Predose and Postdose: 5 minutes; 1; 2; 4; 8; 24; 72 or 96; 144 hours after the end of infusion. Cycle 1 Day 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 7 Day 1: Predose and 5 minutes after the end of infusion
  Time to peak drug concentration in plasma (Tmax)
Pharmacokinetics (PK) of XON7 (Part 2): Tmax | Cycle 1-Day 1; Cycle 2-Day 1; Cycle 3-Day 1; Cycle 6-Day 1; Cycle 9-Day1 and Cycle 12-Day 1: Predose and 5 minutes after the end of infusion
  Time to peak drug concentration in plasma (Tmax)
Pharmacokinetics (PK) of XON7 (Part 1): AUC | Cycle 1-Day 1 Predose and Postdose: 5 minutes; 1; 2; 4; 8; 24; 72 or 96; 144 hours after the end of infusion. Cycle 1 Day 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 7 Day 1: Predose and 5 minutes after the end of infusion
  Area under the plasma concentration versus time curve (AUC). AUC24hours; AUC0-14days and AUC15-28days will be assessed
Pharmacokinetics (PK) of XON7 (Part 2): AUC | Cycle 1-Day 1; Cycle 2-Day 1; Cycle 3-Day 1; Cycle 6-Day 1; Cycle 9-Day1 and Cycle 12-Day 1: Predose and 5 minutes after the end of infusion
  Area under the plasma concentration versus time curve (AUC). AUC24hours; AUC0-14days and AUC15-28days will be assessed
Pharmacokinetics (PK) of XON7 (Part 1): Ctrough | Cycle 1-Day 1 Predose and Postdose: 5 minutes; 1; 2; 4; 8; 24; 72 or 96; 144 hours after the end of infusion. Cycle 1 Day 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 7 Day 1: Predose and 5 minutes after the end of infusion
  Trough concentration (Ctrough) is the concentration reached by XON7 immediately before the next dose is administered
Pharmacokinetics (PK) of XON7 (Part 2): Ctrough | Cycle 1-Day 1; Cycle 2-Day 1; Cycle 3-Day 1; Cycle 6-Day 1; Cycle 9-Day1 and Cycle 12-Day 1: Predose and 5 minutes after the end of infusion
  Trough concentration (Ctrough) is the concentration reached by XON7 immediately before the next dose is administered
Pharmacokinetics (PK) of XON7 (Part 1): Cmin | Cycle 1-Day 1 Predose and Postdose: 5 minutes; 1; 2; 4; 8; 24; 72 or 96; 144 hours after the end of infusion. Cycle 1 Day 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 7 Day 1: Predose and 5 minutes after the end of infusion
  Cmin for the minimum blood plasma concentration reached by XON7 during the time interval between administration of two doses
Pharmacokinetics (PK) of XON7 (Part 2): Cmin | Cycle 1-Day 1; Cycle 2-Day 1; Cycle 3-Day 1; Cycle 6-Day 1; Cycle 9-Day1 and Cycle 12-Day 1: Predose and 5 minutes after the end of infusion
  Cmin for the minimum blood plasma concentration reached by XON7 during the time interval between administration of two doses
Pharmacokinetics (PK) of XON7 (Part 1): T1/2 | Cycle 1-Day 1 Predose and Postdose: 5 minutes; 1; 2; 4; 8; 24; 72 or 96; 144 hours after the end of infusion. Cycle 1 Day 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 7 Day 1: Predose and 5 minutes after the end of infusion
  Half-life (T1/2) refers to the time required for plasma concentration of XON7 to decrease by 50%
Pharmacokinetics (PK) of XON7 (Part 2): T1/2 | Cycle 1-Day 1; Cycle 2-Day 1; Cycle 3-Day 1; Cycle 6-Day 1; Cycle 9-Day1 and Cycle 12-Day 1: Predose and 5 minutes after the end of infusion
  Half-life (T1/2) refers to the time required for plasma concentration of XON7 to decrease by 50%
Pharmacokinetics (PK) of XON7 (Part 1): CL | Cycle 1-Day 1 Predose and Postdose: 5 minutes; 1; 2; 4; 8; 24; 72 or 96; 144 hours after the end of infusion. Cycle 1 Day 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 7 Day 1: Predose and 5 minutes after the end of infusion
  Clearance (CL) is the volume of blood or plasma cleared of XON7 from the body per unit of time
Pharmacokinetics (PK) of XON7 (Part 2): CL | Cycle 1-Day 1; Cycle 2-Day 1; Cycle 3-Day 1; Cycle 6-Day 1; Cycle 9-Day1 and Cycle 12-Day 1: Predose and 5 minutes after the end of infusion
  Clearance (CL) is the volume of blood or plasma cleared of XON7 from the body per unit of time
Pharmacokinetics (PK) of XON7 (Part 1): Vd | Cycle 1-Day 1 Predose and Postdose: 5 minutes; 1; 2; 4; 8; 24; 72 or 96; 144 hours after the end of infusion. Cycle 1 Day 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 7 Day 1: Predose and 5 minutes after the end of infusion
  Volume of distribution (Vd) is defined as the total amount of XON7 in the body divided by its concentration in plasma
Pharmacokinetics (PK) of XON7 (Part 2): Vd | Cycle 1-Day 1; Cycle 2-Day 1; Cycle 3-Day 1; Cycle 6-Day 1; Cycle 9-Day1 and Cycle 12-Day 1: Predose and 5 minutes after the end of infusion
  Volume of distribution (Vd) is defined as the total amount of XON7 in the body divided by its concentration in plasma
Host immunogenicity to XON7 (Part 1 and part 2) | Cycle 1-Day 1; Cycle 1-Day4; Cycle 1-Day7; Cycle 1-Day15; Cycle 2 and additional cycles-Day1; 30 and 60 days after the last dose of XON7
  Number of participants who develop detectable anti-drug antibodies
Host immunogenicity to XON7 (Part 1 and part 2) | Cycle 1-Day 1; Cycle 1-Day4; Cycle 1-Day7; Cycle 1-Day15; Cycle 2 and additional cycles-Day1; 30 and 60 days after the last dose of XON7
  Percentage of participants who develop detectable anti-drug antibodies
Further assess anti-tumor efficacy (Part 1): ORR | Tumor imaging (computed tomography [CT]) will be performed within 28 days prior to enrollment, and while on study approximately every 8 weeks during the treatment period. During the survival follow-up, results of CT only performed in current practice
  Objective response rate (ORR): defined as the proportion of participants with a confirmed complete response [CR] or confirmed partial response [PR] assessed by investigators according to RECIST v1.1. within 3 months after XON7 initiation
Further assess anti-tumor efficacy (Part 2): CBR | Tumor imaging (computed tomography [CT]) will be performed within 28 days prior to enrollment, and while on study approximately every 8 weeks during the treatment period. During the survival follow-up, results of CT only performed in current practice
  Clinical Benefit Rate (CBR) defined as the proportion of participants who achieve CR, PR, and durable SD [SD≥24 weeks] assessed by investigators according to the RECIST criteria v 1.1.
Further assess anti-tumor efficacy (Part 1 and part 2): DCR | Tumor imaging (computed tomography [CT]) will be performed within 28 days prior to enrollment, and while on study approximately every 8 weeks during the treatment period. During the survival follow-up, results of CT only performed in current practice
  Disease control rate (DCR): defined as the proportion of participants who achieve confirmed complete response [CR], confirmed partial response [PR] or stable disease [SD] assessed by investigators according to the RECIST criteria version 1.1.
Further assess anti-tumor efficacy (Part 1 and part 2): DoR | Tumor imaging (computed tomography [CT]) will be performed within 28 days prior to enrollment, and while on study approximately every 8 weeks during the treatment period. During the survival follow-up, results of CT only performed in current practice
  Duration of response (DoR): defined as the time interval between the first confirmed objective response (CR or PR per RECIST 1.1 by investigators) and the first occurrence of objective tumor progression (Progressive disease (PD) per RECIST 1.1 by investigators) or death from any cause.
Further assess anti-tumor efficacy (Part 2): TTR | Tumor imaging (computed tomography [CT]) will be performed within 28 days prior to enrollment, and while on study approximately every 8 weeks during the treatment period. During the survival follow-up, results of CT only performed in current practice
  Time to response (TTR): defined as the time from the date of XON7 initiation to first confirmed objective response (CR or PR per RECIST 1.1 by investigators)..
Further assess anti-tumor efficacy (Part 1 and part 2): PFS | Tumor imaging (computed tomography [CT]) will be performed within 28 days prior to enrollment, and while on study approximately every 8 weeks during the treatment period. During the survival follow-up, results of CT only performed in current practice
  Progression-free survival (PFS): defined as the time from the date of XON7 initiation to the date of first documented progression (RECIST 1.1 by investigators) or death.
Further assess anti-tumor efficacy (Part 1 and part 2): OS | Tumor imaging (computed tomography [CT]) will be performed within 28 days prior to enrollment, and while on study approximately every 8 weeks during the treatment period. During the survival follow-up, results of CT only performed in current practice
  Overall survival (OS): defined as the time interval between the date of XON7 initiation and the date of death due to any cause.
Expansion part: treatment emergent adverse events (TEAEs) | Participants will be assessed for AEs and SAEs beginning immediately after the first dose of investigational drug and continuing through to follow-up which is 60 ± 5 days of last dose of investigational drug.
  An overall summary of AE occurrences with onset during the first treatment cycle will be presented; this will include the following AE attributes:
  * Preferred term,
  * Maximum CTCAE grade,
  * Outcome,
  * Time to first occurrence [days].
Dose Escalation part: clinically significant findings in blood pressure (BP) | Before and immediately after the first dose of investigational drug and continuing through to follow-up which is 60 ± 5 days of last dose of investigational drug
  Incidence and severity of clinically significant findings in blood pressure: Significant blood pressure increase will be defined as BP >150/100 mmHg in a subject without a history of hypertension or increased >20 mmHg (diastolic) from baseline measurement in a subject with a previous history of hypertension.
Dose Escalation part: clinically significant findings in electrocardiogram (ECGs) | Before and immediately after the first dose of investigational drug and continuing through to follow-up which is 60 ± 5 days of last dose of investigational drug
  Incidence of clinically significant findings in Electrocardiogram (ECG): Significant QTc prolongation will be defined as an interval ≥500 msec or an interval which increases by ≥60 msec over baseline
Expansion part: clinically significant changes in Leucocytes count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Leucocytes Count (G/L)
Expansion part: clinically significant changes in Red Blood Cells Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Red Blood Cells Count (T/L)
Expansion part: clinically significant changes in Hemoglobin | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Hemoglobin (g/dL).
Expansion part: clinically significant changes in Hematocrit | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Hematocrit (%).
Expansion part: clinically significant changes in Absolute Neutrophil Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Absolute Neutrophil Count (G/L).
Expansion part: clinically significant changes in Absolute Eosinophil Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Absolute Eosinophil Count (G/L).
Expansion part: clinically significant changes in Absolute Basophil Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Absolute Basophil Count (G/L).
Expansion part: clinically significant changes in Absolute Lymphocytes Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Absolute Lymphocytes Count (G/L).
Expansion part: clinically significant changes in Absolute Monocytes Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Absolute Monocytes Count (G/L).
Expansion part: clinically significant changes in Platelet Count | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Platelet Count (G/L).
Expansion part: clinically significant changes in Albumin | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Albumin (g/L).
Expansion part: clinically significant changes in Bicarbonate | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Bicarbonate (mmol/L).
Expansion part: clinically significant changes in Total Bilirubin | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Total Bilirubin (µmol/L).
Expansion part: clinically significant changes in Calcium | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Calcium (mmol/L).
Expansion part: clinically significant changes in Urea | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Urea (mmol/L).
Expansion part: clinically significant changes in Chloride | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Chloride (mmol/L).
Expansion part: clinically significant changes in Creatinine | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Creatinine (µmol/L).
Expansion part: clinically significant changes in Creatinine Clearance | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Creatinine Clearance (mL/min).
Expansion part: clinically significant changes in Glucose | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Glucose (mmol/L).
Expansion part: clinically significant changes in Magnesium | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Magnesium (mmol/L).
Expansion part: clinically significant changes in Phosphate | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Phosphate (mmol/L).
Expansion part: clinically significant changes in Potassium | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Potassium (mmol/L).
Expansion part: clinically significant changes in Sodium | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Sodium (mmol/L).
Expansion part: clinically significant changes in Total Protein | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Total Protein (g/L).
Expansion part: clinically significant changes in Alanine aminotransferase (ALT) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Alanine aminotransferase (ALT) (U/L).
Expansion part: clinically significant changes in Aspartate aminotransferase (AST) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Aspartate aminotransferase (AST) (U/L).
Expansion part: clinically significant changes in Gamma-glutamyl transférase (GGT) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Gamma-glutamyl transférase (GGT) (U/L).
Expansion part: clinically significant changes in Alkaline Phosphatase (ALP) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Alkaline Phosphatase (ALP) (U/L).
Expansion part: clinically significant changes in Lactate dehydrogenase (LDH) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Lactate dehydrogenase (LDH) (U/L).
Expansion part: clinically significant changes in Amylase | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Amylase (U/L).
Expansion part: clinically significant changes in Lipase | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Lipase (U/L).
Expansion part: clinically significant changes in Total Protein Creatine Kinase (CK) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Total Protein Creatine Kinase (CK) (U/L).
Expansion part: clinically significant changes in Creatine kinase - cardiac muscle isoenzyme (CK-MB) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Creatine kinase - cardiac muscle isoenzyme (CK-MB) (U/L).
Expansion part: clinically significant changes in Troponin T | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Troponin T (ng/L).
Expansion part: clinically significant changes in Prothrombin Time (PT) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Prothrombin Time (PT) (Sec).
Expansion part: clinically significant changes in INR (if under VKA Therapy) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in INR (if under VKA Therapy)
Expansion part: clinically significant changes in Activated Partial Thromboplastin Time (aPTT) | At the end of Cycle 1 (28 days)
  Incidence and magnitude of clinically significant changes in Activated Partial Thromboplastin Time (aPTT) (Sec).

CONTACTS AND LOCATIONS:
Overall Officials: Jaafar BENNOUNA, MD, Principal Investigator — Hôpital Foch
Locations (5):
- Institut Jules Bordet, Anderlecht, Belgium
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Hôpital Foch, Suresnes
  - IUCT-Oncopole, Toulouse